CLINICAL TRIAL: NCT00823017
Title: The Effect of Patient-Preferred Music, Relaxation Music, and Standard Care Environment on Patients in Intensive Care Units
Brief Title: Effect of Music on Patients in Intensive Care Units
Acronym: MTS2
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study withdrawn from IRB
Sponsor: MetroHealth Medical Center (Other)
Collaborators: The Cleveland Music School Settlement (Other); Kulas Foundation (Other); Arthur Flagler Fultz Research Award (American Music Therapy Association) (Unknown)
Responsible Party: Principal Investigator, Charles J. Yowler MD, Professor, Case Western Reserve University School of Medicine, MetroHealth Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB06-00070
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Intensive Care Unit
Keywords: ICU environment; Auditory stimulation; Properties of relaxation music; music; music therapy; pain; anxiety; cortisol; IgA; biomarkers; relaxation music
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Patient-preferred music
  Interventions: Other: Patient-preferred music
- 2 (Experimental): Relaxation Music
  Interventions: Other: Relaxation Music
- 3 (Placebo Comparator): Standard of Care
  Interventions: Other: Standard Care Environment

INTERVENTIONS:
Other: Patient-preferred music — Music of patients' preference
  Arms: 1
Other: Relaxation Music — Relaxation music compiled from results of first three stages of study
  Arms: 2
Other: Standard Care Environment — Control, no interventions
  Arms: 3

SUMMARY:
The purpose of this study is to investigate the effects of patient-preferred music, relaxation music, and standard care environment on patients in intensive care units.

DETAILED DESCRIPTION:
This study is a prospective randomized clinical trial. The purpose of this 4-stage study is to explore the effects of patient-preferred music, relaxation music, and standard care environment on patients in intensive care units.

Stage 1: Recommendation of relaxation music by music therapists who serves as expert panel

Stage 2: Analysis of recommended relaxation music by music therapists

Stage 3: Content validation of relaxation music by healthy adults

Stage 4: Comparison of patients' physiological, psychological, and biological responses to patient-preferred music, relaxation music, and standard care environment

ELIGIBILITY:
Inclusion Criteria:

Communicative (non-intubated, non-sedated)

* At least three days of admission (excluding day of admission)
* 18 years or older
* Mean arterial blood pressure equal or greater than 65 throughout study
* Mean SpO2 equal or greater than 90 throughout study
* Glasgow coma scale equal or greater than 14
* Bilirubin level less than 5
* Ammonia level less than 1
* Hematocrit level greater than 15
* BUN equal or less than 100

Non-communicative (intubated, sedated)

* At least three days of admission (excluding day of admission)
* 18 years or older
* Mean arterial blood pressure equal or greater than 65 throughout study
* Mean SpO2 equal or greater than 90 throughout study
* Glasgow coma scale equal or greater than 10
* Bilirubin level less than 5
* Ammonia level less than 1
* Hematocrit level greater than 15
* BUN equal or less than 100

Exclusion Criteria:

Communicative (non-intubated, non-sedated)

* Patients admitted for or less than 3 days
* Patients with hearing impairments
* Patients with neurological impairments that might impair their ability to process information
* Patients on glucocorticoid medications
* Patients with mental health diagnoses and currently experiencing active psychosis such as hallucinations and/or delusions
* Patient's condition altered dramatically over the 3 days of research

Non-communicative (intubated, sedated)

* Patients admitted for or less than 3 days
* Patients with hearing impairments
* Patients with neurological impairments that might impair their ability to process information
* Patients on glucocorticoid medications
* Patients with mental health diagnoses and currently experiencing active psychosis such as hallucinations and/or delusions
* Patient's condition altered dramatically over the 3 days of research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2010-07 (Actual); Study Completion 2011-03-02 (Actual)

PRIMARY OUTCOMES:
Pain level | 4 data points throughout 1-hour intervention
Anxiety level | 4 data points throughout 1-hour intervention
Comfort level | 4 data points throughout 1-hour intervention
Heart rate | 4 data points throughout 1-hour intervention
Respiration rate | 4 data points throughout 1-hour intervention
Blood pressure | 4 data points throughout 1-hour intervention
Saliva/Serum Cortisol level | 3 data points throughout 1-hour intervention
Saliva/Serum Immunoglobulin A Concentration | 3 data points throughout 1-hour intervention

SECONDARY OUTCOMES:
Psychophysical properties of relaxation music | 1 rating

CONTACTS AND LOCATIONS:
Overall Officials: Xueli Tan, MM, MT-BC, Study Chair — The Cleveland Music School Settlement; Richard B Fratianne, MD, FACS, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States